CLINICAL TRIAL: NCT06481722
Title: Does Knee Joint Angle Affect Muscle Architecture in Children With Spastic Cerebral Palsy?
Brief Title: Knee Joint Angle Affect Muscle Architecture in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, associate professor of pediatric physiotherapy, cairo university, Cairo University
Other Study IDs: P.T.REC/012/ 004995
Record Dates: First submitted 2024-06-22; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Spastic Cerebral Palsy
Keywords: muscle architecture; knee joint angle; cerebral palsy; spasticity; children
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cerebral palsy — no intervention

SUMMARY:
To determine if there is an effect of knee joint angle on muscle architecture in children with spastic cerebral palsy

DETAILED DESCRIPTION:
To determine if there is an effect of knee joint angle on muscle architecture in children with spastic cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of spastic diplegia CP.
* Age from 3 to 6 years.
* Spasticity grade 1 and 1+ according to the Modified Ashworth scale.
* Level III motor function according to the Growth Motor Function Classification System.
* Hamstring muscle tightness.
* Able to understand and follow instructions.

Exclusion Criteria:

* Epilepsy.
* Significant visual or auditory problems according to medical reports (audio-vestibular and ophthalmic examination).
* Structural or fixed soft tissue deformities of the lower extremities.
* Neurological or orthopedic surgery in the past 12 months.
* Botox injection in the lower extremities in the past 6 months.

Ages: 3 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: To determine if there is an effect of knee joint angle on muscle architecture in children with spastic cerebral palsy, 40 diplegic cerebral palsy children of both sexes will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Fascicle length | 3 months
  Fascicle length will be measured by ultrasonography
knee joint angle will be measured by digital Goniometer | 3 months
  knee joint angle will be measured by digital Goniometer
pennation angle | 3 months
  pennation angle will be measured by ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa S Ali, Giza, Married, Egypt

IPD SHARING:
Plan to Share IPD: No